CLINICAL TRIAL: NCT06082453
Title: Modernizing Perinatal Syphilis Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Irene Stafford, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-21-0731; R01HD108201 (NIH)
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis | interventions — Multicenter Studies as Topic; Centers for Disease Control and Prevention, U.S.

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Molecular testing for detection of T. pallidum and use of CDC guidelines for diagnosis of syphilis (Experimental)
  Interventions: Diagnostic Test: Quantitative polymerase chain reaction (qPCR) assay for detection of Treponema pallidum; Diagnostic Test: Aptima Treponema pallidum transcription-mediated amplification (TMA) assay for detection of Treponema pallidum; Other: Center for Disease Control (CDC) Sexually Transmitted Infections (STI) 2021 Treatment Guidelines for diagnosis of syphilis

INTERVENTIONS:
Diagnostic Test: Quantitative polymerase chain reaction (qPCR) assay for detection of Treponema pallidum — A quantitative polymerase chain reaction (qPCR) assay detects and quantifies DNA in a sample, and the qPCR assay used in this study targets the polA gene of T. pallidum to confirm presence of T. pallidum in a sample. Samples will be collected from the mother/newborn dyad at the time of birth. qPCR data will only be used to determine testing performance and will not be used in clinical management of study participants.
Diagnostic Test: Aptima Treponema pallidum transcription-mediated amplification (TMA) assay for detection of Treponema pallidum — The Aptima transcription-mediated amplification (TMA) assay used in this study will target RNA of T. pallidum to confirm presence of T. pallidum in a sample. Samples will be collected from the mother/newborn dyad at the time of birth. TMA data will only be used to determine testing performance and will not be used in clinical management of study participants.
Other: Center for Disease Control (CDC) Sexually Transmitted Infections (STI) 2021 Treatment Guidelines for diagnosis of syphilis — Using the Center for Disease Control (CDC) Sexually Transmitted Infections (STI) 2021 Treatment Guidelines, new born syphilis infection is categorized by clinical providers at birth as follows: confirmed proven/highly probably, possible congenital syphilis (CS), CS less likely, or CS unlikely. These CS categories are determined using neonatal nontreponemal test results, physical exam of the infant, placental pathology, and maternal serologies and treatment history, and comparison of maternal and neonatal nontreponemal tiers. These data will be collected as part of standard clinical care.

SUMMARY:
The purpose of this study is to determine the testing performance of real-time quantitative polymerase chain reaction and transcription mediated amplification by comparing test performance of these novel molecular tests to current 2021 CDC CS guidelines for maternal/neonatal dyads at risk for syphilis infection and to determine whether CS is associated with adverse neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Maternal diagnosis of syphilis by 2021 CDC STI guidelines, irrespective of treatment status; AND viable pregnancy with gestational age ≥ 12 weeks OR postpartum ≤ 96 hours from delivery OR Neonates of pregnancies affected by syphilis ≤ 72 hours of birth
* Individuals (men and non-pregnant) with syphilis in Harris Health clinic with syphilis

Exclusion Criteria:

* Pregnant individuals and neonates who do not meet the criteria of syphilis (false positive)
* Planning to move outside of study prior to ND testing

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 924 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of quantitative polymerase chain reaction (qPCR) assay for detecting T. pallidum | from the time of birth up to 96 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Specificity of quantitative polymerase chain reaction (qPCR) assay for detecting T. pallidum | from the time of birth up to 72 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Positive predictive value of quantitative polymerase chain reaction (qPCR) assay for detecting T. pallidum | from the time of birth up to 72 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Negative predictive value of quantitative polymerase chain reaction (qPCR) assay for detecting T. pallidum | from the time of birth up to 72 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Area under the receiver operating characteristic (ROC) curve of quantitative polymerase chain reaction (qPCR) assay for detecting T. pallidum | from the time of birth up to 72 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Sensitivity of Aptima Treponema pallidum transcription-mediated amplification (TMA) assay for detecting T. pallidum | from the time of birth up to 72 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Specificity of Aptima Treponema pallidum transcription-mediated amplification (TMA) assay for detecting T. pallidum | from the time of birth up to 72 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Positive predictive value of Aptima Treponema pallidum transcription-mediated amplification (TMA) assay for detecting T. pallidum | from the time of birth up to 72 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Negative predictive value of Aptima Treponema pallidum transcription-mediated amplification (TMA) assay for detecting T. pallidum | from the time of birth up to 72 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Area under the receiver operating characteristic (ROC) curve of Aptima Treponema pallidum transcription-mediated amplification (TMA) assay for detecting T. pallidum | from the time of birth up to 72 hours after birth
  Samples will be collected from participants during the following time periods:
  from the time of birth to up to 72 hours after birth (for neonates) from time of birth up to 96 hours after birth (for mothers)
Sensitivity of CDC 2021 STI Treatment Guidelines for diagnosis of syphilis | from 12 weeks gestational age up to 18 months after birth
  Clinical data used to diagnose syphilis according the CDC 2021 STI Guidelines will be collected as part of standard clinical care from the time of pregnancy (greater than or equal to 12 weeks gestational age) up to 18 months after birth.
Specificity of CDC 2021 STI Treatment Guidelines for diagnosis of syphilis | from 12 weeks gestational age up to 18 months after birth
  Clinical data used to diagnose syphilis according the CDC 2021 STI Guidelines will be collected as part of standard clinical care from the time of pregnancy (greater than or equal to 12 weeks gestational age) up to 18 months after birth.
Positive predictive value of CDC 2021 STI Treatment Guidelines for diagnosis of syphilis | from 12 weeks gestational age up to 18 months after birth
  Clinical data used to diagnose syphilis according the CDC 2021 STI Guidelines will be collected as part of standard clinical care from the time of pregnancy (greater than or equal to 12 weeks gestational age) up to 18 months after birth.
Negative predictive value of CDC 2021 STI Treatment Guidelines for diagnosis of syphilis | from 12 weeks gestational age up to 18 months after birth
  Clinical data used to diagnose syphilis according the CDC 2021 STI Guidelines will be collected as part of standard clinical care from the time of pregnancy (greater than or equal to 12 weeks gestational age) up to 18 months after birth.
Area under the receiver operating characteristic (ROC) curve of CDC 2021 STI Treatment Guidelines for diagnosis of syphilis | from 12 weeks gestational age up to 18 months after birth
  Clinical data used to diagnose syphilis according the CDC 2021 STI Guidelines will be collected as part of standard clinical care from the time of pregnancy (greater than or equal to 12 weeks gestational age) up to 18 months after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Stafford, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (9):
- United States (9):
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Nationwide Children's Hospital, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Christus Health, Houston, Texas

IPD SHARING:
Plan to Share IPD: No